CLINICAL TRIAL: NCT07294755
Title: The Impact of Intrapleural Block on Postoperative Pain Caused by Drainage Tubes After Thoracoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jingsheng Lou, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301YXM01
Record Dates: First submitted 2025-11-26; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Saline Solution; Drugs, Investigational; Ropivacaine; Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received normal saline via intrapleural instillation.
  Interventions: Drug: normal saline
- Intervention Group 1 (Experimental): Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received either Investigational Drug ① via intrapleural instillation.
  Interventions: Drug: Investigational drug 20 mL of 0.5% ropivacaine
- Intervention Group 2 (Experimental): Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received either Investigational Drug ② via intrapleural instillation.
  Interventions: Drug: 0.5% ropivacaine + 25 mg tetracaine, made up to a total volume of 20 mL

INTERVENTIONS:
Drug: normal saline — Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received normal saline via intrapleural instillation.
  Arms: Control group
Drug: Investigational drug 20 mL of 0.5% ropivacaine — Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received either Investigational Drug ① via intrapleural instillation.
  Arms: Intervention Group 1
Drug: 0.5% ropivacaine + 25 mg tetracaine, made up to a total volume of 20 mL — Subjects were randomly assigned in a 1:1:1 ratio within 0-24 hours prior to the initiation of elective surgery using computer-generated random numbers. After placement of the thoracic drainage tube, they received either Investigational Drug ② via intrapleural instillation.
  Arms: Intervention Group 2

SUMMARY:
the investigators hereby invite participants to participate in a study entitled "The Impact of Intrapleural Block via Thoracoscopic Surgery on Postoperative Pain Caused by Drainage Tubes". This study is an extension of hospital's major clinical research project: "Efficacy and Safety of Perioperative Intrapleural Block with Local Anesthetics for Acute Postoperative Pain in Adult Thoracic and Pulmonary Surgery: A Prospective, Multicenter, Randomized, Open-Label, Positive Parallel-Controlled, Pragmatic Clinical Trial".During breathing and position changes, the postoperative closed thoracic drainage tube continuously rubs against the pleura, causing severe acute pain in patients. This study hypothesizes that analgesia via a single postoperative spray of local anesthetics into the pleural space is effective, and aims pleural space is effective, and aims to investigate whether a single spray of different local anesthetics can alleviate early acute pain caused by postoperative closed thoracic drainage.

This is a pragmatic randomized controlled study. participants have a 1/3 chance of being randomly assigned to Trial Group A, a 1/3 chance to Trial Group B, and a 1/3 chance to the Control Group. If assigned to Trial Group A, participants will receive an intrapleural block with ropivacaine hydrochloride injection; if assigned to Trial Group B, the intrapleural block will contain both ropivacaine hydrochloride injection and tetracaine hydrochloride injection; if assigned to the Control Group, participants will undergo an intrapleural block without any active medications. All three intrapleural block regimens are fully compatible with the overall disease diagnosis and treatment plan and will not exert any differential impact on participants' subsequent treatment. Additionally, participants' other medical procedures and related costs will not be affected in any way.

Before surgery, as well as at 2, 4, 6, 8, 24, 48 and72 hours after surgery, physicians will conduct follow-up assessments. Participants will also need to complete corresponding follow-up questionnaires under the guidance of doctors. These assessments and questionnaires aim to comprehensively evaluate the analgesic efficacy of the medications, the incidence of postoperative depression, anxiety, cognitive impairment, sleep disturbances, delirium, and adverse reactions, while collecting relevant data. No additional fees will be charged for this process.

Participation in this study is entirely voluntary. Participants may refuse to participate or withdraw from the study at any time during the process without providing any reason. This decision will not affect participants' future medical treatment.

If participants decide to withdraw from the study, please notify participants' research physician in advance. To ensure participants' safety, participants may be required to undergo relevant examinations, which are beneficial for protecting participants' health.

If participants decide to participate in this study, participants' participation and personal data collected during the study will be kept strictly confidential. Physicians in charge of the study and other researchers will use participants' medical information for research purposes only. Participants medical records will be accessible exclusively to the research team. Participants identity will remain anonymous, and only the research physicians and members of the research team will have access to participants' assigned study ID.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* American Society of Anesthesiologists (ASA) physical status classification Ⅰ-Ⅲ, and patients undergoing pulmonary resection via video-assisted thoracic surgery (VATS) under general anesthesia;
* Voluntarily signing the informed consent form;(4) Body Mass Index (BMI) ranging from 18 to 25 kg/m².

Exclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status classification >Ⅲ;
* Patients allergic to amide-type local anesthetics;
* Patients with recent intrathoracic infection;
* Patients with a history of previous pulmonary surgery;
* Patients with long-term alcohol abuse or chronic use of sedatives and analgesics;
* Patients with severe hepatic or renal insufficiency;
* Patients refusing to participate in the study;
* Patients unable to complete the Numeric Rating Scale (NRS);
* Patients expected to be admitted to the Intensive Care Unit (ICU) postoperatively;
* Patients with a Mini-Mental State Examination (MMSE) score <18;
* Pregnant or lactating women;
* Patients with a history of chronic pain;
* Patients not requiring indwelling closed thoracic drainage tube postoperatively;
* Patients converted from video-assisted thoracic surgery (VATS) to thoracotomy intraoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) scores for resting, movement, and coughing | immediately after postoperative awakening； 30 minutes after surgery ； 2 hours after surgery ; 4 hours after surgery ; 6 hours after surgery ; 8 hours after surgery ; 1 day after surgery ; 2 day after surgery ; 3 day after surgery .
  Numeric Rating Scale (NRS) scores for resting, movement, and coughing at the following time points: immediately after postoperative awakening, 30 minutes after surgery , 2 hours, 4 hours, 6 hours, 8 hours, 1 day ; 2 day ; 3 day . The lower the pain score, the greater the patient benefit.

SECONDARY OUTCOMES:
Athens insomnia scale | Baseline 1 day after surgery ; 2 day after surgery ; 3 day after surgery.
  Sleep assessment on postoperative days 1-3: Athens Insomnia Scale (AIS) score. Total score range: 0-24.
  * <4: no sleep disturbance
  * 4-6: sleep disturbance
  * >6: clinical insomnia
The duration of intrapleural analgesia | Within 3 days after surgery; before chest tube removal.
  Duration of intrapleural analgesia: the interval from full emergence (first postoperative C-NRS) until the moment C-NRS ≥ 4 or an increase of ≥ 2 points.
  If the initial C-NRS is already ≥ 4, rescue analgesia is administered and the block is considered ineffective.
Hospital Anxiety and Depression Scale (HADS) scores | Baselineand postoperative day 1; postoperative day 2; postoperative day 3.
  Hospital Anxiety and Depression Scale (HADS) scores pre-operatively and on postoperative days 1-3

OTHER OUTCOMES:
Document drug-related adverse events on postoperative | postoperative day 1 ; postoperative day 2 ; postoperative day 3.
  Document drug-related adverse events on postoperative days 1-3: emergence agitation/delirium, nausea and vomiting, dizziness, respiratory depression, number of rescue analgesia requests, pruritus, disorientation, etc.
Number of PICA demand attempts before chest-drain removal. | Within 3 days after surgery; before chest tube removal.
  Number of IV-PCA demand attempts before chest-drain removal.